CLINICAL TRIAL: NCT01577732
Title: Safety and Reactogenicity of GlaxoSmithKline Biologicals' DTPa-IPV/Hib (Infanrix-IPV+HibTM) in Healthy Vietnamese Toddlers
Brief Title: Safety of GSK Biologicals' Infanrix-IPV+HibTM Vaccine in Healthy Vietnamese Toddlers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 115389; 2013-002538-18 (EudraCT Number)
Record Dates: First submitted 2012-04-05; First posted 2012-04-16 (Estimated); Results first posted 2014-05-05 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Acellular Pertussis; Haemophilus Influenzae Type b; Tetanus; Poliomyelitis; Diphtheria; Diphtheria-Tetanus-aPertussis-Poliomyelitis-Haemophilus Influenzae Type b Vaccines
Keywords: booster; Infanrix-IPV+HibTM; DTPa-IPV/Hib; Vietnamese toddlers
MeSH Terms: conditions — Haemophilus Infections; Tetanus; Poliomyelitis; Diphtheria | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

ARMS (1):
- Infanrix-IPV+Hib Group (Experimental): Subjects aged between, and including 12 and 24 months received a single dose of Infanrix-IPV+Hib™. The vaccine was administered intramuscularly in the anterolateral side of the thigh.
  Interventions: Biological: Infanrix-IPV+Hib™

INTERVENTIONS:
Biological: Infanrix-IPV+Hib™ — Single dose administered intramuscularly (IM) into the anterolateral side of the right thigh.

SUMMARY:
This study aims to evaluate the safety and reactogenicity of a booster dose of Infanrix-IPV+Hib™ when administered to healthy Vietnamese toddlers at 12 to 24 months of age who were vaccinated previously against diphtheria, tetanus, and pertussis diseases within their first six months of lives.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that parent(s)/Legally Acceptable Representative(s) [LAR(s)] can and will comply with the requirements of the protocol.
* A male or female between, and including, 12 and 24 months of age at the time of vaccination.
* Written informed consent obtained from the parent(s)/LAR(s) of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Subjects who were primed with three doses of a DTP and polio vaccine in the first 6 months of life, and who have received the last dose of the primary vaccination at least six months before the receipt of study vaccine.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the dose of study vaccine, or planned use during the study period.
* Administration of a vaccine not foreseen by the study protocol, within 30 days prior to the first study visit, or planned administration during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Evidence of previous or intercurrent booster vaccination against diphtheria, tetanus, pertussis, poliomyelitis and/or Hib disease or vaccination.
* History of any neurological disorders or seizures.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness.
* Acute disease and/or fever at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding vaccination or planned administration during the study period.

Ages: 12 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 321 (Actual)
Dates: Start 2012-12-08 (Actual); Primary Completion 2013-04-09 (Actual); Study Completion 2013-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Haiphong, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=4633

REFERENCES:
- [Background] Anh DD, Van Der Meeren O, Karkada N, Assudani D, Yu TW, Han HH. Safety and reactogenicity of the combined diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae type b (DTPa-IPV/Hib) vaccine in healthy Vietnamese toddlers: An open-label, phase III study. Hum Vaccin Immunother. 2016 Mar 3;12(3):655-7. doi: 10.1080/21645515.2015.1084451. PMID 26337197
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 115389 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115389 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115389 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115389 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115389 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115389 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 321 subjects were screened and allocated a subject number for the study, out of which 300 participated in the study and received the study vaccination.
Groups:
- Infanrix-IPV+Hib Group: Subjects aged between, and including 12 and 24 months received a single dose of Infanrix-IPV+Hib. The vaccine was administered intramuscularly in the anterolateral side of the thigh.
Period: Overall Study
Arm/Group | Infanrix-IPV+Hib Group
Started | 300
Completed | 300
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Infanrix-IPV+Hib Group
Number analyzed (Participants) | 300
Age, Continuous [Mean (Standard Deviation); unit: months] | 15.8 (2.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 143
  Male | 157
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - South East Asian Heritage | 300

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Solicited Local Symptoms
Description: Solicited local symptoms assessed were pain, redness and swelling. Any = occurrence of any local symptom regardless of intensity grade.
Time Frame: Within the 4-day (Days 0-3) follow up period after vaccination.
Population: Analyses were performed on the Total Vaccinated cohort, which included all the subjects with documented administration of the study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-IPV+Hib Group
Number analyzed (Participants) | 300
Participants
  Any Pain | 95
  Any Redness | 82
  Any Swelling | 52

2. Primary Outcome: Number of Subjects Reporting Solicited General Symptoms
Description: Solicited general symptoms assessed were Drowsiness, Irritability/Fussiness, Loss of Appetite and Fever, defined as axillary temperature higher than (>) 37.5 degrees Celsius (°C). Any = occurrence of a general symptom regardless of intensity grade or relationship to study vaccination.
Time Frame: Within the 4-day (Days 0-3) follow up period after vaccination.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-IPV+Hib Group
Number analyzed (Participants) | 300
Participants
  Any Drowsiness | 52
  Any Irritability/fussiness | 108
  Any Loss of appetite | 115
  Any Fever | 101

3. Primary Outcome: Number of Subjects Reporting Any Unsolicited Adverse Events (AEs).
Description: An unsolicited AE was any AE (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any = occurrence of an AE regardless of intensity grade or relationship to study vaccination.
Time Frame: Within the 31-day (Days 0-30) follow up period after vaccination.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-IPV+Hib Group
Number analyzed (Participants) | 300
Participants | 107

4. Primary Outcome: Number of Subjects Reporting Any Serious Adverse Events (SAEs).
Description: SAEs assessed included medical occurrences that resulted in death, were life threatening, required hospitalization or prolongation of hospitalization or resulted in disability/incapacity. Any SAE = any SAE regardless of assessment of relationship to study vaccination.
Time Frame: During the entire study period (Days 0-30).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-IPV+Hib Group
Number analyzed (Participants) | 300
Participants | 1

ADVERSE EVENTS:
Time Frame: Solicited symptoms: 4-day (Days 0-3) follow-up period after booster vaccination; unsolicited AEs: 31-day (Days 0-30) follow-up period after booster vaccination; SAEs: during the entire study period (Days 0-30).
Arm/Group | Infanrix-IPV+Hib Group
All-Cause Mortality (participants affected / at risk) | 0/300
Serious Adverse Events (participants affected / at risk) | 1/300
Other Adverse Events (participants affected / at risk) | 211/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infanrix-IPV+Hib Group (N=300)
Convulsion (Nervous system disorders) | 1
Pneumonia (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Infanrix-IPV+Hib Group (N=300)
Pain (General disorders) | 95
Redness (General disorders) | 82
Swelling (General disorders) | 52
Drowsiness (General disorders) | 52
Irritability/fussiness (General disorders) | 108
Loss of appetite (General disorders) | 115
Fever (General disorders) | 101
Cough (Respiratory, thoracic and mediastinal disorders) | 48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.